CLINICAL TRIAL: NCT04279990
Title: Assessment of Gastric Motility on Funtional Dyspepsia and Joint Hypermobility Syndrome
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S56804
Record Dates: First submitted 2020-02-11; First posted 2020-02-21 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Functional Dyspepsia; Joint Hypermobility Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Functional dyspepsia patients with JHS: Patients with functional dyspepsia as defined by the Rome III criteria and joint hypermobility syndrome as defined by the Beighton Hypermobility criteria.
  Interventions: Other: No intervention: assessment of GI function
- Functional dyspepsia patients without JHS: Patients with functional dyspepsia as defined by the Rome III criteria and WITHOUT joint hypermobility syndrome as defined by the Beighton Hypermobility criteria.
  Interventions: Other: No intervention: assessment of GI function
- Healthy subjects: Healthy subjects with no gastrointestinal diseases including no functional dyspepsia
  Interventions: Other: No intervention: assessment of GI function

INTERVENTIONS:
Other: No intervention: assessment of GI function — Gastrointestinal function is assessed by the intragastric pressure measurement by a high resolution manometry. This is an examination test considered standard of care for the diagnosis of functional dyspepsia in the university hospital of leuven.
  The joint hypermobility syndrome is assess by means of the Brighton criteria.
  Other Names: No intervention: assessment of JHS

SUMMARY:
Functional dyspepsia (FD) is defined as the presence of gastroduodenal symptoms in the absence of organic disease that is likely to explain the symptoms. Joint hypermobility (JH) refers to the increased passive or active movement of a joint beyond its normal range. Recent reports have highlighted the co-existence of FD with Ehlers-Danlos syndrome type III or hypermobility type (EDSIII). The association between FD and EDS III, and the underlying pathophysiological alterations, are poorly understood. We hypothesised that EDS III might influence gastroduodenal sensorimotor function, resulting in dyspeptic symptoms. Therefore, the aim of this study is to explore the impact of EDS III on gastric motility, nutrient tolerance and dyspeptic symptoms in patients with functional dyspepsia.Our aim is to study the prevalence of EDSIII in FD compared to healthy subjects (HS) and to study the impact of co-existing EDSIII on gastric motility, nutrient tolerance and dyspeptic symptoms in FD.

ELIGIBILITY:
Inclusion Criteria:

- Patients with PDS diagnosis as per Rome III by Rome III questionnaire

Exclusion Criteria:

Patients are excluded from the study if any of the following criteria are met:

* Females who are pregnant or lactating.
* Patients who are H. Pylori positive
* Patients with confirmed gastro-intestinal disease, with former digestive surgery affecting upper gut motility, a concomitant disease responsible for digestive symptoms
* Patients presenting with predominant symptoms of irritable bowel syndrome (IBS), CIN or GERD.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with PDS diagnosis as per Rome III by Rome III questionnaire and healthy subjects with out gastrointestinal symptoms
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2014-07-04 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Gastric motility in JHS and non-JHS | 2 years
  This is a physiological parameter. Intragastric pressure measurement (mmHg) in JHS and non-JHS are compared to the Intragastric pressure measurement (mmHg) of healthy subjects. During the intragastric pressure measurement, the pressure drop (mmHg) from baseline during the intragastric infussion of a liquid meal will be assessed and compared in both groups (patients vs. controls).
Prevalence of JHS in functional dyspepsia | 2 years
  The number of patients with JHS and without JHS will be assessed. Based on the number of patients in each group, propotions (in %) can be calculated of the presence of JHS in a functional dyspepsia cohort.

SECONDARY OUTCOMES:
Prevalence of dyspepsia symptoms | 2 years
  prevalence of dyspepsia symptoms in FD patients with JHS compared to patients without JHS.
Level of nutrient tolerance during the intragastric pressure measurement in JHS | 2 years
  During the intragastric pressure assessment, a liquid nutrient drink is intragastrically infussed until the subjects experience and repport maximal satiation. Maximal satiation is assessed every minute during the intragastric infussion of the nutrient drink by means of questionnaires (VAS score: 0, no sensation; 5, maximal satiation). For this outcome, the quantity of nutrient drink tolerated during the test will be measured (ml) in patients with and without JHS and compared.
Level of nutrient tolerance during the intragastric pressure measurement in patients vs controls | 2 years
  During the intragastric pressure assessment, a liquid nutrient drink is intragastrically infussed until the subjects experience and repport maximal satiation. Maximal satiation is assessed every minute during the intragastric infussion of the nutrient drink by means of questionnaires (VAS score: 0, no sensation; 5, maximal satiation). For this outcome, the quantity of nutrient drink tolerated during the test will be measured (ml) in patients with and without JHS and will be compared with the amount of volume (ml) assessed in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven

REFERENCES:
- [Derived] Carbone F, Goelen N, Fikree A, Aziz Q, Tack J. Impact of joint hypermobility syndrome on gastric accommodation and nutrient tolerance in functional dyspepsia. Neurogastroenterol Motil. 2021 Jul;33(7):e14086. doi: 10.1111/nmo.14086. Epub 2021 Feb 2. PMID 33528850